CLINICAL TRIAL: NCT02944422
Title: The Prevalence of Oral Habits in a Group of Primary School Children in Cairo Governorate: A Cross-Sectional Study
Brief Title: The Prevalence of Oral Habits in a Group of Primary School Children in Cairo Governorate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Hassan Saad, Dr, Cairo University
Other Study IDs: CEBC-CU-2016-10-142
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Oral Habit

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Males: Primary school Egyptian boys from 7-10 years.
- Females: Primary school Egyptian girls from 7-10 years.

SUMMARY:
This study is designed to determine the prevalence of oral habits among primary Egyptian school children in Cairo Governorate, Egypt.

DETAILED DESCRIPTION:
This aim of this study is to determine the prevalence of oral habits among primary Egyptian school children in Cairo Governorate, Egypt.

PICO:

P: Egyptian primary school children of 7 - 10 years old

O: Prevalence of oral habits

Primary Outcome: Prevalence of Oral Habit; Device of Measurement: Questionnaire; Unit of Measurement: Binary.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children of 7-10 years old
* Children with no intellectual problems

Exclusion Criteria:

* Children with orthodontic appliances
* Medically compromised children
* Children of families who refuse to participate in the study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary school Egyptian children.
Sampling Method: Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Oral Habit | 5 months
  Measurement that will be used: Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hamdy, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shetty SR, Munshi AK. Oral habits in children--a prevalence study. J Indian Soc Pedod Prev Dent. 1998 Jun;16(2):61-6. PMID 11813757
- [Background] Quashie-Williams R, daCosta OO, Isiekwe MC. Oral habits, prevalence and effects on occlusion of 4-15 year old school children in Lagos, Nigeria. Niger Postgrad Med J. 2010 Jun;17(2):113-7. PMID 20539325
- [Background] Onyeaso CO. Oral habits among 7-10 year-old school children in Ibadan, Nigeria. East Afr Med J. 2004 Jan;81(1):16-21. doi: 10.4314/eamj.v81i1.8789. PMID 15080510
- [Background] Lagana G, Masucci C, Fabi F, Bollero P, Cozza P. Prevalence of malocclusions, oral habits and orthodontic treatment need in a 7- to 15-year-old schoolchildren population in Tirana. Prog Orthod. 2013 Jun 14;14:12. doi: 10.1186/2196-1042-14-12. PMID 24326142
- [Background] Kharbanda OP, Sidhu SS, Sundaram K, Shukla DK. Oral habits in school going children of Delhi: a prevalence study. J Indian Soc Pedod Prev Dent. 2003 Sep;21(3):120-4. PMID 14703220
- [Background] M Hegde A, M Xavier A. Childhood Habits: Ignorance is not Bliss- A Prevalence Study. Int J Clin Pediatr Dent. 2009 Jan;2(1):26-9. doi: 10.5005/jp-journals-10005-1037. Epub 2009 Apr 26. PMID 25206095
- [Background] Guaba K, Ashima G, Tewari A, Utreja A. Prevalence of malocclusion and abnormal oral habits in North Indian rural children. J Indian Soc Pedod Prev Dent. 1998 Mar;16(1):26-30. PMID 11813715
- [Background] Garde JB, Suryavanshi RK, Jawale BA, Deshmukh V, Dadhe DP, Suryavanshi MK. An epidemiological study to know the prevalence of deleterious oral habits among 6 to 12 year old children. J Int Oral Health. 2014 Feb;6(1):39-43. Epub 2014 Feb 26. PMID 24653601
- See also: Related Info — http://www.aapd.org/media/policies_guidelines/g_developdentition.pdf
- See also: Related Info — http://www.columbia.edu/itc/hs/dental/d7710/client_edit/oral_habits_slides_printout.pdf